CLINICAL TRIAL: NCT05951608
Title: A Phase Ib/II Open-label Clinical Study to Evaluate the Safety, Tolerability and Preliminary Efficacy of AK127 in Combination With AK112 in Patients With Advanced Malignant Tumors
Brief Title: A Phase Ib/II Clinical Study of AK127 in Combination With AK112 in Patients With Advanced Solid Tumors
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK127-104
Record Dates: First submitted 2023-07-11; First posted 2023-07-19 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AK127 in combination with AK112 (Experimental): Subjects will receive AK127 in combination with AK112 by intravenous administration
  Interventions: Drug: AK127 in combination with AK112

INTERVENTIONS:
Drug: AK127 in combination with AK112 — AK127 in combination with AK112 (administered on Day 1 of each cycle, Q3W) up to 2 years

SUMMARY:
A Phase Ib/II Open-label Clinical Study to Evaluate the Safety, Tolerability and Preliminary Efficacy of AK127 in combination with AK112 in Patients with Advanced Malignant Tumors

DETAILED DESCRIPTION:
The study consisted of two parts. The first part, Phase Ib is to characterize the safety, tolerability, pharmacokinetics (PK), immunogenicity of AK127 in combination with AK112 in adult subjects with advanced solid tumor malignancies. The part, as a dose escalation phase is to determine the maximum tolerated dose (MTD), or recommended Phase 2 dose (RP2D) for AK127 in combination with AK112, and describe Dose Limiting Toxicity (DLT).The second part, Phase II is to Evaluate the anti-tumor activity of AK127 in combination with AK112 in different tumor species cohorts.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and voluntarily sign a written informed consent form (ICF), which must be signed before the specified study procedures required for the study are performed.
2. Males or females aged ≥ 18 to ≤ 75 years at the time of signing informed consent.
3. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0 or 1.
4. Life expectancy ≥3 months；
5. Histologically or cytologically documented advanced or metastatic solid tumor that is refractory/relapsed to standard therapies, or for which no effective standard therapy is available, or the subject is not suitable for standard therapy.
6. Adequate organ function.
7. Patients of childbearing potential must agree to use effective contraceptive measures.

Exclusion Criteria:

1. The patient has received prior immunotherapy against TIGIT target.
2. The patient had previously been treated with anti-PD -(L)1 and anti-VEGF targets.
3. Currently enrolled in any other clinical study.
4. Receipt of any anticancer therapy within 4 weeks prior to the first dose of Investigational drug;
5. Symptomatic central nervous system metastases.
6. Active malignancies within the past 3 years, with the exception of tumors in this study and cured local tumors
7. Active autoimmune disease requiring systemic treatment prior to the start of study treatment.
8. There is a history of major diseases 1 year prior to the first dose.
9. Medical history of gastrointestinal perforation or gastrointestinal fistula within 6 months prior to the first dose
10. Received chest radiation therapy prior to the first dose
11. Presence of clinically symptomatic pleural effusion, pericardial effusion, or ascites requiring frequent drainage.
12. Active or previously documented inflammatory bowel disease (e.g., Crohn's disease or ulcerative colitis).
13. Receipt of live or attenuated vaccination within 4 weeks prior to the first dose of Investigational drug.
14. Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
15. Known history of active tuberculosis.
16. History of organ transplant or hematopoietic stem cell.
17. History of primary immunodeficiency.
18. Any condition that, in the opinion of the investigator, would interfere with evaluation of the investigational product or interpretation of subject safety or study results.
19. Other cases deemed inappropriate by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2023-07 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) | From the subject signs the ICF to 30 days (AE) and 90 days (SAE) after the last dose of study treatment or initiation of other anti-tumor therapy, whichever occurs first
  An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product temporally associated with the use of study treatment, whether or not considered related to the study treatment
Number of participants with a Dose Limiting Toxicity (DLT) | During the first 3 weeks
  DLTs will be assessed during the first 3 weeks of treatment for dose-escalation Ib phase and are defined as toxicities that meet pre-defined severity criteria, and assessed as having a suspected relationship to study drug, and unrelated to disease, disease progression, inter-current illness, or concomitant medications that occurs within the first cycle (3 weeks) of treatment
Number of participants with ORR | Up to 2 years
  Efficacy measures such as overall response rate (ORR), which is the proportion of subjects with CR or PR by investigator based on RECIST v1.1
Progression-Free Survival | Up to 2 years
  PFS is defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurs first assessed by investigator Per RECIST 1.1.

SECONDARY OUTCOMES:
Disease control rate | Up to 2 years
  DCR, which is defined as the proportion of subjects with CR, PR, or SD, based on RECIST v1.1
Duration of response | Up to 2 years
  DoR, which is defined as the duration from the first documentation of objective response to the first documented disease progression or death due to any cause, whichever occurs first.
Time to Progress | Up to 2 years
  TTR is defined as the time to response base on RECIST v1.1
AUC of AK127 and AK112 | Up to 2 years
  Area under the curve (AUC) of AK127 and AK112
PK of AK127 and AK112 | Up to 2 years
  The endpoints for assessment of PK of AK127 and AK112 include serum concentrations of AK127 and AK112 at different timepoints after AK127 and AK112 administration
Cmax of AK127 and AK112 | Up to 2 years
  Maximum observed concentration (Cmax) of AK127 and AK112
Cmin of AK127 and AK112 at steady state | Up to 2 years
  Minimum observed concentration (Cmin) of AK127 and AK112 at steady state
The immunogenicity of AK127 and AK112 | Up to 2 years
  The immunogenicity of AK127 and AK112 will be assessed by summarizing the number of subjects who develop detectable anti-drug antibodies (ADAs)

CONTACTS AND LOCATIONS:
Overall Officials: shun lu, MD, Principal Investigator — Shanghai Chest Hospital; yun fan, MD, Principal Investigator — Zhejiang Cancer Hospital